CLINICAL TRIAL: NCT06048614
Title: The Administration of Saline Enema Versus Glycerin Suppository as a Treatment Intervention for Meconium Obstruction of Prematurity (MOP) and to Study the Impact on the Resolution of MOP, Time to Reach Full Enteral Feeds, Gut Microbiome, and Gut-brain Axis, a Randomised Control Trial.
Brief Title: Saline Enema Administration in Meconium Obstruction of Prematurity and Impact on the Resolution, Feeds, Microbiome, and Gut-brain Axis.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Collaborators: Singapore General Hospital (Other); Genome Institute of Singapore (Other); Translational Immunology Institute (Unknown); Duke-NUS Graduate Medical School (Other)
Responsible Party: Principal Investigator, Thowfique Kadavukarayil Ibrahim, Senior Consultant(Assistant Professor), KK Women's and Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023/2270
Record Dates: First submitted 2023-08-03; First posted 2023-09-21 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Meconium Obstruction of Prematurity
MeSH Terms: conditions — Meconium Ileus

STUDY DESIGN:
Intervention Model Description: The treatment group will receive SE with normal saline (20-40 ml/kg/per SE) 2 times a day at 48 to 72 hrs of age at the earliest. The infant with medical instability procedure will be deferred until the infant is medically fit and intervention is continued until the infant reaches full feeds, defined as 110 ml/kg/day or yellow stools whichever is earlier. SE will be recommenced if the infant does not open bowel for 2 days before reaching full feeds. In ≤ 750 grams infant, paediatric surgeons would perform the first catheterisation with 6F catheter, insertion length will be limited to 8 cm, and saline is infused with the aid of gravity. Syringe flushing is allowed if gravity force fail to drive saline to the intestine.Two ultrasound abdominal examination will be performed and first scan will coincide with first SE in 500-750 grams infants.Failure to resolve the MOP with SE will be designated as treatment failure and managed with contrast enema or Laparotomy by paediatric surgeons.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Saline Enema Arm) (Experimental): After randomisation, infant who allocated with intervention group will proceed with SE with normal saline (20-40ml/kg twice daily) earliest at 48 to 72 hours of age. Then continue until 2 days of yellow stools/ 110ml/kg/day of oral feeds; whichever is earlier.
  SE are recommended if baby do not do bowel opening (BO) for 2 days before reaching full feeds
  Interventions: Procedure: Saline Enema (SE)
- Control Arm (Glycerin Suppository Arm) (Active Comparator): Infants randomized to GS received the standard management protocol for meconium retention in the unit. GS (2,000 mg, a quarter unit, four doses 12 h apart) were administered to infants earliest at 48 hour to 72 hours of birth, with subsequent once-daily GS being administered at the discretion of the managing team. Infants who were diagnosed with meconium obstruction later in the first 2 weeks of life were also treated with glycerin suppositories for 48 hrs, with subsequent once-daily GS being administered at the discretion of the managing team.
  Infants who failed to respond to glycerin suppositories were referred to the surgical team by the managing team The subsequent management of meconium retention was at the surgeon's discretion and included continued GS by the surgical team, contrast enema or surgical interventions performed in escalating order as mentioned.
  Interventions: Drug: Glycerin Suppository

INTERVENTIONS:
Procedure: Saline Enema (SE) — infant who allocated with intervention group will proceed with SE with normal saline (20-40ml/kg twice daily) at 48 hours of age. Then continue until 2 days of yellow stools/ 110ml/kg/day of oral feeds; whichever is earlier.
  SE are recommended if baby do not do bowel opening (BO) for 2 days before reaching full feeds
  Failure to resolve the MOP with SE will be designated as treatment failure and managed with contrast enema or Laparotomy by paediatric surgeons, following a formal referral.GS is not allowed in intervention arm
  Arms: Intervention Arm (Saline Enema Arm)
Drug: Glycerin Suppository — Infants randomized to GS received the standard management protocol for meconium retention in the unit. GS (2,000 mg, a quarter unit, four doses 12 h apart) were administered to infants earliest at 48 hour to 72 hours of birth, with subsequent once-daily GS being administered at the discretion of the managing team. Infants who were diagnosed with meconium obstruction later in the first 2 weeks of life were also treated with glycerin suppositories for 48 hrs, with subsequent once-daily GS being administered at the discretion of the managing team.
  Infants who failed to respond to glycerin suppositories were referred to the surgical team by the managing team The subsequent management of meconium retention was at the surgeon's discretion and included continued GS by the surgical team, contrast enema or surgical interventions performed in escalating order as mentioned.
  Arms: Control Arm (Glycerin Suppository Arm)

SUMMARY:
The goal of this clinical trial is to study the effect of twice-daily saline enema (SE) in the treatment obstruction of prematurity (MOP) in infants with the birth weight ≤1.25kg. The main questions, the trial aims to answer are

1. To validate the finding of our pilot study which had shown that twice-daily SE reduces the time to reach full enteral feeds in premature infant as compared to premature infant treated with Glycerine Suppository (GS), in a larger cohort. Infant with MOP fails to pass meconium in the first 48 hours of life and develop symptoms and signs like abdominal distension and feed intolerance.
2. The other aims of this study are to test whether the intervention is

   1. Effective treatment for MOP
   2. Reduce the duration of ICU stay
   3. Reduce the rate of necrotizing enterocolitis, sepsis, Total Parenteral Nutrition (TPN) days and number of intravenous catheter days
3. The study also wants to explore the impact of this intervention on the gut microbiome, gut-brain interaction and immune response of the new-born.

DETAILED DESCRIPTION:
Very low birth weight infants (VLBW ≤ 1.5 kg) constitute more than 60% of bed occupancy in level III neonatal units. They face the risk of 10-50% long-term disability, and their initial healthcare cost ranges from S$50,000 to 1 million, an important healthcare issue.

The incidence of meconium obstruction of prematurity (MOP) is 20-30% in extremely low birth weight (ELBW ≤ 1 kg) infants. The intervention based on the current standard of care increase the risk of laparotomy necrotizing enterocolitis, intestinal perforation, and neurodevelopmental risks posed by general anaesthesia. Our published pilot RCT demonstrated that saline enema (SE) is an effective, feasible, and safe intervention to reduce the time to reach full enteral feeds and is a potentially effective treatment for MOP in ELBW (< 1 kg) infants.

Our primary hypothesis is that Infants with Twice-daily high-volume SE (20-40 ml/kg/day) intervention will result in reduced time to reach full enteral feeds compared to infants treated with conventional management with Glycerin suppository (GS) in (≤1.25kg) infants with MOP. Our exploratory hypothesis is that SE will have a protective effect on the gut microbiome, inflammatory and immune response in preterm infants.

Ninety-five infants born over three years in KK Hospital (KKH) and Singapore General Hospital (SGH) will be enrolled and randomized at 48 hours or later to receive SE or GS. The standardized protocol will be used for the accreditation and administration of SE. Primary, secondary, and exploratory outcomes data, including treatment failure data, will be recorded. Infants will be followed up to 36 weeks of gestation or discharge, whichever is earlier. Maternal and infant characteristics, inflammatory and immune response, and safety outcome data will be collected.

If the findings of our pilot trial are confirmed, the protocol can become the standard of care in preterm infants with MOP. Additionally, significant healthcare cost savings will be realized alongside an improved understanding of the Microbiome, immune and inflammatory response pertaining to the gut.

ELIGIBILITY:
Inclusion Criteria:

* Criteria A: For infant presenting with early onset of MOP

  1. Birth weight 500 - 1250 gram
  2. ≥ 23 weeks gestation
  3. No BO for 48 hours
  4. BO present but with a small amount or stain of meconium
  5. Feeds intolerance or abdominal X-ray showing dilated loops of bowel
* Criteria B: For infant presenting with Late onset of MOP

  1. Birth weight 500 - 1250 gram
  2. ≥ 23 weeks gestation
  3. Infants who passed meconium initially and develop evidence of meconium obstruction at a later age (feed intolerance or vomiting and abnormal abdominal X-ray with or without abdominal distension)

Exclusion Criteria:

Infants that:

1. Neuromuscular disorder
2. Moderate or severe asphyxia
3. Inability to start enteral feeding, which continued for 3 consecutive days before 2 weeks of post-natal age for reasons unrelated to meconium inspissation or its complication
4. Without parental consent
5. Aggravated medical instability
6. Single mothers < 21 years

Ages: 1 Day to 36 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 95 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to reach full enteral feeds in days | Before 36 weeks of corrected age of discharge of the infant
  Time to reach full enteral feeds is measured from birth to the time infant reaches full oral milk feeds.
  Full oral milk feed is defined as milk volume of 110ml/kg/day. The total parenteral nutrition is discontinued when infant reaches milk feed volume of 110ml/kg/day.
  Rationale:
  SE loosens the thick and sticky meconium by saline absorption and triggers effective and strong peristaltic contractions, thereby leading to the evacuation of meconium from the gut. The evacuation of meconium leads to the resolution of the gut obstruction, thereby enhancing feed tolerance in premature infants with meconium obstruction of prematurity.

SECONDARY OUTCOMES:
Rate of treatment failure | Before 36 weeks of corrected age of discharge of the infant
  Treatment failure is defined as the need to use additional treatment measures, apart from the study intervention to resolve MOP in the study cohort.
Rate of (a) Culture positive sepsis (b) Necrotising enterocolitis. | Before 36 weeks of corrected age of discharge of the infant
  Rationale:
  If twice daily SE leads to the shortening of time to reach full enteral feeds, resolution of MOP, and promote friendly bacteria microbiome, then it has the potential to reduce NICU stay, risk of necrotising enterocolitis, risk of sepsis, duration of total parenteral nutrition, duration of PICC and overall cost of care.
Duration in days of (a) ICU stay (b) Total parenteral nutrition (c) PICC days. | Before 36 weeks of corrected age of discharge of the infant
  Rationale:
  If twice daily SE leads to the shortening of time to reach full enteral feeds, resolution of MOP, and promote friendly bacteria microbiome, then it has the potential to reduce NICU stay, risk of necrotising enterocolitis, risk of sepsis, duration of total parenteral nutrition, duration of PICC and overall cost of care.
Overall cost of care calculated in SGD at the time of discharge | Before 36 weeks of corrected age of discharge of the infant
  Rationale:
  If twice daily SE leads to the shortening of time to reach full enteral feeds, resolution of MOP, and promote friendly bacteria microbiome, then it has the potential to reduce NICU stay, risk of necrotising enterocolitis, risk of sepsis, duration of total parenteral nutrition, duration of PICC and overall cost of care.

OTHER OUTCOMES:
Identification and quantification of bacteria from meconium/stool samples by DNA sequencing and analysis of top 50 bacteria Genus | Before 36 weeks of corrected age of discharge of the infant
  Bacteria are identified from meconium/stools samples, collected at birth and weekly interval till discharge or 36 weeks of gestation
To measure the serum level of IL 6 in pg/ml | Before 36 weeks of corrected age of discharge of the infant
  Use Olink Target 48 platform to measure
  Rationale:
  To explore the relationship between gut microbiome and gut-brain axis
To measure the serum level of neurotransmitters noradrenaline in pg/L | Before 36 weeks of corrected age of discharge of the infant
  Use Norepinephrine ELISA Kit from abcam to measure
Measure serum levels of dopamine in arbitrary units (peak area of analyte divided by peak area of an internal standard) | Before 36 weeks of corrected age of discharge of the infant
  Use Norepinephrine ELISA Kit from abcam to measure
Measure serum levels of serotonin in arbitrary units (peak area of analyte divided by peak area of an internal standard) | Before 36 weeks of corrected age of discharge of the infant
  Use Norepinephrine ELISA Kit from abcam to measure
Measure serum levels of GABA in arbitrary units (peak area of analyte divided by peak area of an internal standard) | Before 36 weeks of corrected age of discharge of the infant
  Use Norepinephrine ELISA Kit from abcam to measure
Measure level of Propionate in µM | Before 36 weeks of corrected age of discharge of the infant
  Use Short Chain Fatty Acid Panel to measure
Measure level of Butyrate in µM | Before 36 weeks of corrected age of discharge of the infant
  Use Short Chain Fatty Acid Panel to measure
Measure level of Acetate in µM | Before 36 weeks of corrected age of discharge of the infant
  Use Short Chain Fatty Acid Panel to measure

CONTACTS AND LOCATIONS:
Overall Officials: Thowfique Ibrahim, FRCPCH, FAMS, Principal Investigator — Singhealth Duke-NUS Medical School, NUS and LKC Medical School
Locations (2):
- Singapore (2):
  - Singapore General Hospital, Singapore
  - KK Women's and Children Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Unger A, Goetzman BW, Chan C, Lyons AB 3rd, Miller MF. Nutritional practices and outcome of extremely premature infants. Am J Dis Child. 1986 Oct;140(10):1027-33. doi: 10.1001/archpedi.1986.02140240073029. PMID 3092638
- [Background] Chathas MK, Paton JB, Fisher DE. Percutaneous central venous catheterization. Three years' experience in a neonatal intensive care unit. Am J Dis Child. 1990 Nov;144(11):1246-50. doi: 10.1001/archpedi.1990.02150350078030. PMID 2239866
- [Background] Stoll BJ, Gordon T, Korones SB, Shankaran S, Tyson JE, Bauer CR, Fanaroff AA, Lemons JA, Donovan EF, Oh W, Stevenson DK, Ehrenkranz RA, Papile LA, Verter J, Wright LL. Late-onset sepsis in very low birth weight neonates: a report from the National Institute of Child Health and Human Development Neonatal Research Network. J Pediatr. 1996 Jul;129(1):63-71. doi: 10.1016/s0022-3476(96)70191-9. PMID 8757564
- [Background] Shim SY, Kim HS, Kim DH, Kim EK, Son DW, Kim BI, Choi JH. Induction of early meconium evacuation promotes feeding tolerance in very low birth weight infants. Neonatology. 2007;92(1):67-72. doi: 10.1159/000100804. Epub 2007 Mar 14. PMID 17356305
- [Background] Krasna IH, Rosenfeld D, Salerno P. Is it necrotizing enterocolitis, microcolon of prematurity, or delayed meconium plug? A dilemma in the tiny premature infant. J Pediatr Surg. 1996 Jun;31(6):855-8. doi: 10.1016/s0022-3468(96)90153-0. PMID 8783123
- [Background] Emil S, Nguyen T, Sills J, Padilla G. Meconium obstruction in extremely low-birth-weight neonates: guidelines for diagnosis and management. J Pediatr Surg. 2004 May;39(5):731-7. doi: 10.1016/j.jpedsurg.2004.01.027. PMID 15137008
- [Background] Haiden N, Norooz F, Klebermass-Schrehof K, Horak AS, Jilma B, Berger A, Repa A. The effect of an osmotic contrast agent on complete meconium evacuation in preterm infants. Pediatrics. 2012 Dec;130(6):e1600-6. doi: 10.1542/peds.2011-3634. Epub 2012 Nov 26. PMID 23184118
- [Background] Broussard DL. Gastrointestinal motility in the neonate. Clin Perinatol. 1995 Mar;22(1):37-59. PMID 7781255
- [Background] Dumont RC, Rudolph CD. Development of gastrointestinal motility in the infant and child. Gastroenterol Clin North Am. 1994 Dec;23(4):655-71. PMID 7698826
- [Background] Campbell BG, Couceyro P, Keana JF, Weber E. N-methyl-D-aspartate receptor-mediated contractions of the guinea pig ileum longitudinal muscle/myenteric plexus preparation: modulation by phencyclidine and glycine receptors. J Pharmacol Exp Ther. 1991 May;257(2):754-66. PMID 1674535
- [Background] Siddiqui MM, Drewett M, Burge DM. Meconium obstruction of prematurity. Arch Dis Child Fetal Neonatal Ed. 2012 Mar;97(2):F147-50. doi: 10.1136/adc.2010.190157. Epub 2010 Nov 29. PMID 21115553
- [Background] Juang D, Snyder CL. Neonatal bowel obstruction. Surg Clin North Am. 2012 Jun;92(3):685-711, ix-x. doi: 10.1016/j.suc.2012.03.008. Epub 2012 Apr 17. PMID 22595716
- [Background] Kim YJ, Kim EK, Kim ES, Kim HS, Choi JH, Cheon JE, Kim WS, Kim IO, Park KW. Recognition, diagnosis and treatment of meconium obstruction in extremely low birth weight infants. Neonatology. 2012;101(3):172-8. doi: 10.1159/000330850. Epub 2011 Oct 22. PMID 22024741
- [Background] Garza-Cox S, Keeney SE, Angel CA, Thompson LL, Swischuk LE. Meconium obstruction in the very low birth weight premature infant. Pediatrics. 2004 Jul;114(1):285-90. doi: 10.1542/peds.114.1.285. PMID 15231948
- [Background] Cho HH, Cheon JE, Choi YH, Lee SM, Kim WS, Kim IO, Shin SM, Kim EK, Kim HS, Choi JH, You SK. Ultrasound-guided contrast enema for meconium obstruction in very low birth weight infants: Factors that affect treatment success. Eur J Radiol. 2015 Oct;84(10):2024-31. doi: 10.1016/j.ejrad.2015.06.006. Epub 2015 Jun 7. PMID 26159485
- [Background] Ibrahim T, Li Wei C, Bautista D, Sriram B, Xiangzhen Fay L, Rajadurai VS. Saline Enemas versus Glycerin Suppositories to Promote Enteral Feeding in Premature Infants: A Pilot Randomized Controlled Trial. Neonatology. 2017;112(4):347-353. doi: 10.1159/000477999. Epub 2017 Aug 3. PMID 28768263
- [Background] Paradiso VF, Briganti V, Oriolo L, Coletta R, Calisti A. Meconium obstruction in absence of cystic fibrosis in low birth weight infants: an emerging challenge from increasing survival. Ital J Pediatr. 2011 Nov 14;37:55. doi: 10.1186/1824-7288-37-55. PMID 22082231
- [Background] Livingston MH, Shawyer AC, Rosenbaum PL, Williams C, Jones SA, Walton JM. Glycerin enemas and suppositories in premature infants: a meta-analysis. Pediatrics. 2015 Jun;135(6):1093-106. doi: 10.1542/peds.2015-0143. Epub 2015 May 18. PMID 25986027
- [Background] Vinson AE, Houck CS. Neurotoxicity of Anesthesia in Children: Prevention and Treatment. Curr Treat Options Neurol. 2018 Oct 13;20(12):51. doi: 10.1007/s11940-018-0536-z. PMID 30315440
- [Background] Saenz de Pipaon Marcos M, Teresa Montes Bueno M, Sanjose B, Gil M, Parada I, Amo P. Randomized controlled trial of prophylactic rectal stimulation and enemas on stooling patterns in extremely low birth weight infants. J Perinatol. 2013 Nov;33(11):858-60. doi: 10.1038/jp.2013.86. Epub 2013 Aug 1. PMID 23907087
- [Background] Nakaoka T, Nishimoto S, Tsukazaki Y, Santo K, Higashio A, Kamiyama M, Uehara S, Yoneda A, Tanaka Y, Ichiba H. Ultrasound-guided hydrostatic enema for meconium obstruction in extremely low birth weight infants: a preliminary report. Pediatr Surg Int. 2017 Sep;33(9):1019-1022. doi: 10.1007/s00383-017-4129-9. Epub 2017 Jul 25. PMID 28744798